CLINICAL TRIAL: NCT02174523
Title: Pharmacokinetic Study of Lurasidone After Multiple Oral Administration in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Collaborators: Xuhui Central Hospital, Shanghai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D1070003
Record Dates: First submitted 2014-02-11; First posted 2014-06-25 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2014-06

CONDITIONS: Schizophrenia
Keywords: pharmacokinetic; lurasidone; multiple dose
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 40mg lurasidone (Experimental): Single oral administration of 40 mg study drug lurasidone after the over 350 kcal breakfast on Day 1. Administration was suspended on Days 2 and 3. Continuous oral administration of 40 mg study drug lurasidone, once daily between Day 4 and Day 8.
  Interventions: Drug: 40mg lurasidone
- placebo (Placebo Comparator): Single oral administration of 40 mg study drug placebo after the over 350 kcal breakfast on Day 1. Administration was suspended on Days 2 and 3. Continuous oral administration of 40 mg placebo, once daily between Day 4 and Day 8.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 40mg lurasidone
  Arms: 40mg lurasidone
Drug: placebo
  Arms: placebo

SUMMARY:
To evaluate the pharmacokinetic (PK) characteristics after multiple oral administration of 40 mg lurasidone in healthy Chinese subjects.

To evaluate the safety and tolerance after multiple oral administration of 40 mg lurasidone in healthy Chinese subjects.

DETAILED DESCRIPTION:
Single oral administration of 40 mg study drug lurasidone or placebo after the over 350 kcal breakfast on Day 1. Administration was suspended on Days 2 and 3. Continuous oral administration of 40 mg study drug lurasidone or placebo, once daily between Day 4 and Day 8.

ELIGIBILITY:
Inclusion Criteria:

1. After detailed explanations of study objectives, methods and procedures, anticipated efficacy, pharmacologic actions, risks and other relevant contents, subjects are aware of all relevant information related to this study and have signed the informed consent form voluntarily.
2. Male subjects are 18≤ age <40 years of age when signing the informed consent.
3. Subjects with body weight of 50.0≤ and ≤80.0 kg and BMI (body mass index) of 19.0≤ and <24.0 at screening examination.
4. Subjects are able to comply with all requirements during this study period, receive various physical and laboratory examinations per study protocol, and report subjective symptoms.

Exclusion Criteria:

1. Based on the examination results during screening period, various physical and laboratory examinations performed 1 day before medication (Day -1) and before administration of study drug on the medication day, there are certain medical concerns on subject's health status in principal investigator's or study supervising physician's opinions (certain treatment or medical observation are deemed necessary).
2. Subjects with past diabetic history.
3. Subjects has an HbA1c level of >6.2% at screening.
4. Subjects with history of gastrointestinal operations (excluding appendectomy).
5. Because of subjects' past medical history of cardiovascular diseases, liver diseases, renal diseases, endocrine disorders, digestive diseases, hematologic diseases, respiratory diseases, mental illness, neurological disorders (especially epilepsy and other convulsive disorders) and other diseases, subjects are unsuitable to participate in this study in the principal investigator's or study supervising physician's opinions.
6. Subjects with past history of allergy to drugs.
7. Subjects have consumed grapefruit or food containing grapefruit ingredients between 7 days before medication (Day_-7) and before administration of study drug on the medication day (Day 1). Subjects have consumed food containing hypericum perforatum L. ingredients between 14 days before medication (Day_-14) and administration of study drug on the medication day (Day 1).
8. Subjects have taken any drugs (including over-the-counter drugs) between 7 days before medication (Day_-7) and before administration of study drug on medication day.
9. Regular drinker (criteria are mean daily consumption ≥2 bottles of 640 mL beers or Chinese liquor≥150 mL).
10. Subjects are used to drink large amount (criteria are daily consumption>1.8 L) of caffeine-containing beverages (e.g. coffee, black tea, green tea, coca cola or nutritional oral solution, etc).
11. Subjects have history of drug abuse or positive urine drug tests.
12. Subjects with positive immunologic test results.
13. Average amount of daily smoking>20 cigarettes.
14. Subjects have taken other study drugs within 3 months (Day_-90~Day 1) before medication.
15. Subjects received lurasidone orally before.
16. Subjects have history of blood donations of 400 mL within 3 months (Day_-90~Day 1) before medication; 200 mL within 1 month (Day_-30~Day 1) before medication; or donation of blood components within 2 weeks (Day_-14~Day 1) before medication.
17. Subjects have consumed alcohol-containing food between 3 days before medication 3 (Day_-3) and before administration of study drug on medication day.
18. Subjects can not tolerate venipuncture or have poor peripheral venous access.
19. Subjects are unwilling to abstain from vigorous exercise from Day_-1 until discharge.
20. Other subjects who are unsuitable to participate in this study in principal investigator's or study supervising physician's opinions.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ChaoYing Hu, MD, Principal Investigator — Xuhui Center Hospital, Shanghai
Locations (1):
- Xuhui Center Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hu C, Wang Y, Song R, Yu C, Luo X, Jia J. Single- and Multiple-Dose Pharmacokinetics, Safety and Tolerability of Lurasidone in Healthy Chinese Subjects. Clin Drug Investig. 2017 Sep;37(9):861-871. doi: 10.1007/s40261-017-0546-8. PMID 28695535

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 27 subjects were screened at the clinical site after obtaining informed consent. A total 14 subjects were enrolled into the study and were randomized to lurasidone group (10) and placebo group (4). The data of informed consent from the first subject was 8th April 2014（and that from the last subject was 15th April 2014）.
Period: Overall Study
Arm/Group | 40mg Lurasidone | Placebo
Started | 10 | 4
Completed | 9 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received lurasidone or placebo were included in the safety population. All subjects who received lurasidone and have evaluable PK data were included in the PK analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | 40mg Lurasidone | Placebo | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (3.74) | 26.5 (5.07) | 27.4 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Lurasidone Cmax
Description: Maximum (peak) observed drug serum concentration.
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
ng/mL | 50.2 (44.3)

2. Primary Outcome: Lurasidone AUC 0-24
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
ng･h/mL | 152 (33.2)

3. Primary Outcome: Lurasidone AUC 0-τ
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
ng･h/mL | 166 (32.4)

4. Primary Outcome: Lurasidone AUC0-∞
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Standard Deviation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
ng･h/mL | 179 (29.9)

5. Primary Outcome: Lurasidone Tmax
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Median (Full Range); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
h | 1.50 [1.0 to 4.0]

6. Primary Outcome: Lurasidone λz
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
1/h | 0.0360 (20.8)

7. Primary Outcome: Lurasidone t1/2
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
h | 19.3 (20.8)

8. Primary Outcome: Lurasidone MRT
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
h | 12.2 (22.7)

9. Primary Outcome: Lurasidone CL/F
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
L/h | 223 (29.9)

10. Primary Outcome: CLss/F
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
L/h | 211 (27.9)

11. Primary Outcome: Lurasidone Vz/F
Time Frame: pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
L | 6198 (47.9)

12. Primary Outcome: Lurasidone Vzss/F
Time Frame: Day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
L | 10618 (38.6)

13. Primary Outcome: Accumulation Ratios Lurasidone,Ratio of Cmax,Ratio of AUC0-∞,Ratio of AUC0-τ,
Time Frame: Day 8/Day 1
Measure: Mean (90% Confidence Interval); unit: Ratios
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
Ratios
  Ratio of Cmax | 0.94 [0.75 to 1.18]
  Ratio of AUC0-∞ | 1.74 [1.59 to 1.90]
  Ratio of AUC0-τ | 1.25 [1.14 to 1.36]
  Ratio of Cτ | 2.52 [2.37 to 2.68]

14. Primary Outcome: Summary of Concentration (ng/mL) of Lurasidone - PK Population the Mean (SD) of Day 4 and Day 5
Time Frame: Pre-dose (-0.5h) of Day4 and Day5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 10
ng/ml
  Day4 Pre-dose (-0.5h) | 0.277 (31.5)
  Day5Pre-dose (-0.5h) | 1.15 (28.7)

15. Primary Outcome: Summary of Concentration (ng/mL) of Lurasidone - PK Population the Mean (SD) of Day 6 and Day 7
Time Frame: Pre-dose (-0.5h) of Day6 and Day7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 9
ng/ml
  Day6 Pre-dose (-0.5h) | 1.56 (27.1)
  Day7 Pre-dose (-0.5h) | 2.00 (27.3)

16. Primary Outcome: Lurasidone Cmax
Description: Maximum (peak) observed drug serum concentration.
Time Frame: Day8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
ng/mL | 48.5 (49.4)

17. Primary Outcome: Lurasidone AUC 0-24
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
ng･h/mL | 190 (27.9)

18. Primary Outcome: Lurasidone AUC 0-τ
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
ng･h/mL | 234 (27.4)

19. Primary Outcome: Lurasidone AUC0-∞
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng･h/mL
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
ng･h/mL | 314 (26.6)

20. Primary Outcome: Lurasidone Tmax
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Median (Full Range); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
h | 1.75 [1.0 to 4.0]

21. Primary Outcome: Lurasidone λz
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
1/h | 0.0199 (20.2)

22. Primary Outcome: Lurasidone t1/2
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
h | 34.9 (20.2)

23. Primary Outcome: Lurasidone MRT
Time Frame: Day8 0.5hours pre-dose, 0.5,1,1.5,2,3,4,6,8,12,24,36,48 hours post-dose in day 8
Population: All subjects with evaluable PK data were included in PK data analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | 40mg Lurasidone
Number analyzed (Participants) | 8
h | 22.0 (19)

ADVERSE EVENTS:
Arm/Group | 40mg Lurasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 10/10 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40mg Lurasidone (N=10) | Placebo (N=4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood prolactin increased (Investigations) | 6 (6) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 10 (10) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Restlessness (Psychiatric disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other